CLINICAL TRIAL: NCT00088829
Title: A Pilot Study to Establish a Standardized Protocol for Gene Microarray Analysis in Patients Receiving Neoadjuvant Chemotherapy for Breast Cancer: Identifying Factors Predictive of a Response to Paclitaxel
Brief Title: Genetic Testing in Predicting Response to Paclitaxel in Women With Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Investigator left institution
Sponsor: Georgetown University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CDR0000368453; P50CA058185 (NIH); P30CA051008 (NIH); GUMC-00310
Record Dates: First submitted 2004-08-04; First posted 2004-08-05 (Estimated); Results first posted 2018-07-11 (Actual); Last update posted 2018-07-11 (Actual); Status verified 2018-05

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; stage IA breast cancer; stage IB breast cancer; HER2-negative breast cancer; HER2-positive breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel; Microarray Analysis; Biopsy; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Paclitaxel (Experimental): Paclitaxel given before surgery
  Interventions: Drug: paclitaxel; Genetic: microarray analysis; Procedure: biopsy; Procedure: neoadjuvant therapy

INTERVENTIONS:
Drug: paclitaxel — subjects will receive paclitaxel neoadjuvantly
Genetic: microarray analysis — subjects will have a biopsy to collect tissue for gene microarray analysis
Procedure: biopsy — All subjects will have a biopsy to collect tissue
Procedure: neoadjuvant therapy — paclitaxel is given neoadjuvantly
Drug: Paclitaxel — All patients will receive paclitaxel neoadjuvantly
  Other Names: Taxol

SUMMARY:
RATIONALE: Analyzing genes for changes before and after chemotherapy may help doctors predict a patient's response to treatment and help plan the most effective treatment.

PURPOSE: This clinical trial is studying how well genetic testing works in predicting response to paclitaxel in women who have unresected breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the feasibility of accruing women with unresected infiltrating carcinoma of the breast to a clinical trial involving serial breast biopsies and administration of neoadjuvant paclitaxel before formal assessment of axillary lymph node status.
* Determine a standard protocol template for gene microarray analysis, in terms of the timing and method of collecting tissue samples, before and after administration of neoadjuvant paclitaxel in these patients.
* Determine the safety and efficacy of tissue sampling in these patients.

Secondary

* Identify gene(s) or gene clusters that exhibit significant differences between responding and non-responding tumors before treatment with neoadjuvant paclitaxel in these patients.
* Identify gene(s) or gene clusters that exhibit changes in gene expression before and after the administration of neoadjuvant paclitaxel in these patients.
* Compare significant differences in gene expression between responding and non-responding tumors in patients treated with this drug.
* Develop, preliminarily, a statistical model utilizing individual genes and/or gene clusters that can best predict response to paclitaxel in these patients.

OUTLINE: This is a pilot, multicenter study.

Patients undergo core needle breast biopsy within 14 days before starting neoadjuvant paclitaxel treatment. Patients receive neoadjuvant paclitaxel IV over 3 hours on day 1. Treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.

Patients undergo core needle breast biopsy 48 hours after the first administration of paclitaxel, upon completion of course 1, and either upon completion of the last course (in patients with clinical or radiographic evidence of residual disease) or during definitive breast surgery. Biopsy samples are analyzed for gene expression by gene microarray analysis.

Patients are followed for survival.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study within 2 years.

ELIGIBILITY:
Inclusion:

* Histologically confirmed infiltrating carcinoma of the breast

  * Unresected disease
  * High-risk (> 50% risk of relapse) disease, including any of the following high-risk markers:

    * Estrogen receptor- and progesterone receptor- negative
    * Palpable axillary lymph nodes
    * Grade 3 histology
    * S phase fraction > 10%
    * Ki67 > 30%
* Disease that warrants combination therapy with doxorubicin, cyclophosphamide, and paclitaxel
* HER2/neu negative or positive
* Hormone receptor status:

  * Not specified

Menopausal status

* Known

Performance status

* ECOG 0-2
* Absolute neutrophil count > 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Bilirubin ≤ 1. 5 times normal (except for patients with known Gilbert's disease)
* Creatinine ≤ 1.5 times normal

Exclusion:

* uncontrolled congestive heart failure
* myocardial infarction within the past 6 months
* unstable angina
* uncontrolled hypertension
* pregnant or nursing
* serious bacterial, viral, or fungal infection requiring ongoing treatment
* severe peripheral neuropathy
* poor psychiatric risk
* history of any other known serious co-morbid medical or psychiatric condition
* prior cytotoxic therapy for breast cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2001-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Minetta C. Liu, MD, Principal Investigator — Lombardi Comprehensive Cancer Center
Locations (1):
- Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Paclitaxel
Started | 22
Completed | 0
Not Completed | 22
Not completed — PI left institution and study was close | 22

BASELINE CHARACTERISTICS:
Arm/Group | Paclitaxel
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Overall Response
Description: Due to the early termination of the study, this data for this outcome was not collected.
Time Frame: 3 months
Arm/Group | Paclitaxel
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: Due to the early termination of the study, no adverse event data was recorded.
Arm/Group | Paclitaxel
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes